CLINICAL TRIAL: NCT05255250
Title: PLAYshop: A Parent-focused Physical Literacy Intervention for Early Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Victoria (Other); Women and Children's Health Research Institute (WCHRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PLAYshop2022
Record Dates: First submitted 2022-01-10; First posted 2022-02-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Motor Activity; Parent-Child Relations; Child Development
Keywords: Questionnaires; Interviews; Fundamental movement skill assessments; Accelerometers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will complete baseline measures and then be randomly assigned to group 1 (intervention) or group 2 (control), in a computer generated1:1 sequence.
Who Masked: Participant
Masking Description: Participants: While the families will not be told explicitly if they have been assigned to the intervention or control group, they may be able to determine their group based on when their workshop is scheduled (i.e., immediately versus after completion of all study measures).
  Research Coordinator: The research coordinator will be aware of the group allocations as they will be in charge of coordinating random assignment and have to schedule participants into workshops and other measures based on their specific allocation.
  Outcomes Assessors: Research assistants who score children's fundamental movement skills based on recorded videos will not be told explicitly if a participant is part of the intervention or control group. Though there is a possibility that they may recall group assignment from previous data collection sessions they led.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLAYshop Intervention (Experimental): Participants will receive a 60 minute virtual physical literacy workshop, an equipment goody-bag with basic play equipment and printed resources, and access to a digital app with an online toolkit and four bi-weekly boosters lessons.
  Interventions: Behavioral: PLAYshop
- Control (No Intervention): Participants will receive the 60 minute virtual physical literacy workshop, equipment goody-bag, and access to the digital app after completing 2-month follow-up measures.

INTERVENTIONS:
Behavioral: PLAYshop — The intervention includes: 1. Educational Training - the 60 min virtual workshop will be delivered by a trained facilitator. Parents will be introduced to physical literacy via education, group discussion, and active participation in fundamental movement skills (FMS) based activities with their child. 2. Distribution of Education Resources- Parents will be sent physical literacy and physical activity printed resources. 3. Material resources -parents will also be provided a bag of inexpensive active play equipment (e.g., ball, bean bag, balloons). 4. Provide Follow-up Support- After the workshop, participants will gain access to an app with an online toolkit including new active play ideas, tips, and equipment they can make at home for active play. Additionally, participants will receive four bi-weekly booster lessons that include key workshop messages, support and encouragement for parents, reflection and check-in questions, and new activities to try with their child.
  Arms: PLAYshop Intervention

SUMMARY:
The PLAYshop program is a novel, brief, theory-based, parent-focused physical literacy intervention designed to address this major public health issue of childhood physical inactivity and to support families.

Primary Research Question: Does the PLAYshop program increase preschool-aged children's physical literacy, including fundamental movement skills and motivation and enjoyment, compared to controls?

DETAILED DESCRIPTION:
The overall goal for the proposed study is to examine the efficacy of the PLAYshop program, a novel, brief, theory-based, parent-focused physical literacy intervention, on child- and family-specific outcomes.

Research Questions:

Primary: Does the PLAYshop program increase preschool-aged children's physical literacy, including fundamental movement skills and motivation and enjoyment, compared to controls? Secondary: Does the PLAYshop program increase preschool-aged children's physical activity and co-participation in physical activity with parents, compared to controls? Tertiary: 1) Does the PLAYshop program increase parents' capability, motivation, and opportunity to support preschool-aged children's physical literacy development, compared to controls? 2) What is the level of, and factors that influence, implementation at the family and program delivery level?

Hypotheses:

Increases in preschool-aged children's fundamental movement skills, motivation and enjoyment, physical activity, and parent-child co-participation in physical activity will be greater in the intervention group, compared to the control group. Additionally, increase in parents' capability, motivation, and opportunity to support preschool-aged children's physical literacy development will be greater in the intervention group, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-5 years and their parents
* Living in non-rural areas of Alberta or British Columbia, Canada as defined by Statistics Canada

Exclusion Criteria:

* Children diagnosed with developmental delay or disorder/condition that may affect gross motor development or limit their ability to be physically active.
* Families with parents who do not comfortably speak or read English.
* Families that do not have access to a smartphone/tablet with camera and microphone.
* Families that have participated in prior PLAYshop pilot and feasibility trials.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in children's physical literacy (fundamental movement skills) | Baseline and 2 month follow-up
  Children's fundamental movement skills, including two manipulative skills (i.e., overhand throw, underhand throw), two locomotor skills (i.e., horizontal jump, hop), and one balance/stability skill (i.e., one leg balance), will be assessed in a recorded virtual meeting. The skills are from the Test of Gross Motor Development (TGMD) and the Movement Assessment Battery for Children-Second Edition (MABC-2).
Change in children's physical literacy (motivation and enjoyment; parental report) | Baseline and 2 month follow-up
  Children's motivation and enjoyment will be assessed via a parental questionnaire that includes items from the Preschool Physical Literacy Assessment (Pre PLAy). This scale includes 4 items with values of 1-5; higher values mean more motivation and enjoyment. Citation: Cairney et al. (2018)
Change in children's physical literacy (enjoyment; child report) | Baseline and 2 month follow-up
  Children's enjoyment will also be assessed via self-report using an adapted Five Degrees of Happiness Likert scale for children. This scale includes 1 item with a value of 1-5; a higher value means more enjoyment. Citation: Hall et al. (2016)

SECONDARY OUTCOMES:
Change in children's physical activity | Baseline and 2 month follow-up
  Children's physical activity will be assessed with Actigraph wGT3X-BT accelerometers worn for 7 consecutive days. Validated cut-points for preschool-aged children will be used to classify each 15 second count into sedentary time or physical activity.
Change in parent-child co-participation in physical activity (accelerometer) | Baseline and 2 month follow-up
  Parent-child co-participation in physical activity will be assessed with Actigraph wGT3X-BT accelerometers worn for 7 consecutive days by children and designated parents. Validated cut-points for preschool-aged children and adults will be used to classify each 15 second count into sedentary time or physical activity. The Bluetooth proximity detection feature on the accelerometer will be enabled to determine the presence (e.g., same room in a house, at the park together) or absence of close proximity between two accelerometers.
Change in parent-child co-participation in physical activity (questionnaire) | Baseline and 2 month follow-up
  Parent-child co-participation in physical activity will also be assessed with a parental questionnaire. This scale includes 4 items with values of 1-5; higher values mean more co-participation in PA. Citation: Mâsse et al., 2020
Change in parental physical activity modelling | Baseline and 2 month follow-up
  Parental physical activity modelling will be assess via a parental questionnaire. This scale includes 3 items with values of 1-4: higher values mean higher modelling. Citation: Davison et al., 2011

OTHER OUTCOMES:
Change in parents' capability to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop, approximately 1-2 weeks after baseline (intervention), one week after baseline (control), 2-month follow-up (all)
  Parental capability (i.e., knowledge), will be assessed via a parental questionnaire. This scale includes 9 items with values of 1-5; higher values mean more capability.
Change in parents' motivation to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop, approximately 1-2 weeks after baseline (intervention), one week after baseline (control), 2-month follow-up (all)
  Parental motivation (i.e., confidence (11 items), beliefs (4 items), outcome expectations (3 items), intentions (2 items), perceived behavioural control (4 items)) will be assessed via a parental questionnaire. Citation for beliefs and outcome expectations: Heitzler et al., 2006. Items have values of 1-5; higher values mean more parental motivation.
Change in parents' opportunity to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop, approximately 1-2 weeks after baseline (intervention), one week after baseline (control), 2-month follow-up (all)
  Parental opportunity (e.g., perceived availability of resources (1 item), perceived barriers (5 items)) will be assessed via a parental questionnaire. Items have values of 1-5; higher values mean less parental opportunity. Citation for perceived barriers: Heitzler et al., 2006
Implementation: satisfaction and perceived usefulness (questionnaire) | Intervention group: Immediately after the workshop
  Satisfaction and perceived usefulness of the intervention will be assessed via a parental questionnaire in the intervention group only. This scale includes 3 items with values of 1-5; higher values mean more satisfaction and perceived usefulness.
Implementation: satisfaction and perceived usefulness (parental interview) | Intervention group: 2-month follow-up
  Satisfaction and perceived usefulness of the intervention will also be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: facilitators and barriers (parental interview) | Intervention group: 2-month follow-up
  Implementation facilitators and barriers will be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: facilitators and barriers (workshop leader interview) | At study completion, approximately 1 year from first workshop.
  Implementation facilitators and barriers will be explored via brief semi-structured interviews with workshop leaders.
Implementation: dose (parental interview) | Intervention group: 2-month follow-up
  The dose of the intervention will be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: dose (app check-in questions) | Intervention group: Bi-weekly after workshop (i.e., 1, 3, 5, and 7 weeks)
  The dose of the intervention will be assessed via check-in questions as part of the booster lessons in the intervention group.
Implementation: dose (app usage data) | Intervention group: 2-month follow-up
  The dose of the intervention will be assessed via tracking of app usage in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Carson, PhD, Principal Investigator — University of Alberta; Patti-Jean Naylor, PhD, Principal Investigator — University of Victoria; Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Sam Liu, PhD, Principal Investigator — University of Victoria
Locations (1):
- Kinesiology, Sport, and Recreation, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
To protect participant's personal data, IPD will not be shared with researchers outside of the research team.

REFERENCES:
- [Background] Masse LC, O'Connor TM, Lin Y, Carbert NS, Hughes SO, Baranowski T, Beauchamp MR. The physical activity parenting practices (PAPP) item Bank: a psychometrically validated tool for improving the measurement of physical activity parenting practices of parents of 5-12-year-old children. Int J Behav Nutr Phys Act. 2020 Nov 4;17(1):134. doi: 10.1186/s12966-020-01036-0. PMID 33148276
- [Background] Heitzler CD, Martin SL, Duke J, Huhman M. Correlates of physical activity in a national sample of children aged 9-13 years. Prev Med. 2006 Apr;42(4):254-60. doi: 10.1016/j.ypmed.2006.01.010. Epub 2006 Feb 20. PMID 16490241
- [Background] Hall, L., Hume, C., & Tazzyman, S. (2016). Five Degrees of Happiness: Effective Smiley Face Likert Scales for Evaluating with Children. In Proceedings of the The 15th International Conference on Interaction Design and Children (311-321). ACM.
- [Background] Cairney J, Clark HJ, James ME, Mitchell D, Dudley DA, Kriellaars D. The Preschool Physical Literacy Assessment Tool: Testing a New Physical Literacy Tool for the Early Years. Front Pediatr. 2018 Jun 7;6:138. doi: 10.3389/fped.2018.00138. eCollection 2018. PMID 29930933
- [Background] Davison KK, Li K, Baskin ML, Cox T, Affuso O. Measuring parental support for children's physical activity in white and African American parents: the Activity Support Scale for Multiple Groups (ACTS-MG). Prev Med. 2011 Jan;52(1):39-43. doi: 10.1016/j.ypmed.2010.11.008. Epub 2010 Nov 25. PMID 21111755
- [Derived] Carson V, Boyd M, Potter M, Rhodes R, Liu S, Naylor PJ. Protocol for the PLAYshop randomised controlled trial: examining efficacy of a virtually delivered parent-focused physical literacy intervention for early childhood on child-specific and family-specific outcomes. BMJ Open. 2022 Dec 22;12(12):e066962. doi: 10.1136/bmjopen-2022-066962. PMID 36549741